CLINICAL TRIAL: NCT06356363
Title: Development of a Questionnaire on Patients' Perception of Their Oncology Care Pathway
Brief Title: Development of a Questionnaire on Patients' Perception of Their Oncology Care Pathway (Onco-PREMs)
Acronym: OncoPREMs
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Jean-Godinot (Other)
Collaborators: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_005_OncoPREMs
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Oncology; oncology care pathway; patients' perception; questionnaire; psychometric validation
MeSH Terms: conditions — Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patient: Patient with cancer regardless of location or stage.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — data collection

SUMMARY:
Healthcare systems are evolving, giving increasing prominence to the patient-centered model, accompanied by objective and perceived outcomes.

PREMs (Patient Reported Experience Measures) are used to assess how patients feel about their experience of care. PREMs enable patients to take an active role in their own care, and enable healthcare establishments to identify areas for improvement that can be incorporated into their quality processes.

In oncology, the collection of patient-perceived quality regarding their care pathway would enable better coordination of their care. While a few initiatives have emerged in the field of PREMs, the development of a reliable questionnaire assessing patient perception of their care pathway in oncology remains a challenge.

DETAILED DESCRIPTION:
The aims of the study are to constitute a questionnaire to assess patients' perceptions of their oncology care pathway and to perform its psychometric validation.

ELIGIBILITY:
Inclusion Criteria:

* cancer patient
* regardless of location or stage
* Fluent in French
* aged more than 18 years old
* Agreeing to take part in the study

Exclusion Criteria:

* With an estimated life expectancy of less than 3 months
* In remission, untreated or without follow-up for more than 12 months
* Protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cancer regardless of location or stage.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Psychometric validation | Day 0
  Stastistical analysis to confirm the psychometric validation of the IGQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: DIOURI Loubna, Principal Investigator — Institut Godinot

IPD SHARING:
Plan to Share IPD: Undecided